CLINICAL TRIAL: NCT06048263
Title: The Perinatal SMILES (Synergistic Multi-component Intervention to alLeviate dEpressive Symptoms) Case Series. Combining Ketamine and Interpersonal Psychotherapy to Improve Postpartum Mood
Brief Title: The Perinatal Synergistic Multi-component Intervention to alLeviate dEpressive Symptoms. A Case Series
Acronym: SMILES
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: PI is leaving the university
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, David Monks, Assoc Prof of Anesthesiology, Anesthesiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202306156
Record Dates: First submitted 2023-08-15; First posted 2023-09-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Postpartum Depression
Keywords: Pregnancy; Socio-economically disadvantaged; Cesarean; Postpartum depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Interpersonal Psychotherapy; adenylate isopentenyltransferase; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Interpersonal psychotherapy plus ketamine (Experimental): Five sessions of interpersonal psychotherapy (IPT) and pre-, and post-, ketamine sessions b) Two doses of subcutaneous (SC) ketamine in the first 4 post-cesarean days
  Interventions: Behavioral: interpersonal psychotherapy (IPT); Drug: Ketamine

INTERVENTIONS:
Behavioral: interpersonal psychotherapy (IPT) — The ROSE intervention is a five-session intervention developed to build communication skills, improve social support, and improve stress management. It is easy to learn and does not require a healthcare professional or mental health specialist to deliver. For this study, the investigators plan to deliver to individuals during inpatient visits, in-person appointments or via telemedicine (phone or videoconference), as appropriate or per participant preference. The first four sessions are approximately 60 minutes in length.
  Other Names: Reach Out Stay Strong Essentials (ROSE) IPT
Drug: Ketamine — During the first four post-cesarean days, the investigators will administer subcutaneous ketamine (0.5 mg/kg) and a repeated dose of 0.5 or 0.7 mg/kg ~24 hours later (the second dose will be increased to 0.7 mg/kg if no severe adverse effects are reported after the first dose and the patient is in agreement with the dose escalation).
  Other Names: Subcutaneous Ketamine

SUMMARY:
The goal of this open label case series is to learn about the feasibility of conducting a future randomised controlled trial to evaluate how well the Perinatal SMILES intervention works in improving post-cesarean mood in low-income women.

The main questions it aims to answer are:

1. Is it feasible to recruit a sufficient number of participants?
2. Is it feasible to administer Perinatal SMILES and
3. Is it feasible to collect participant outcomes?

To profile EEG in participants at rest and in response to TMS, before and after subcutaneous ketamine

Participants will:

1. Complete five sessions of interpersonal therapy
2. Receive two skin injections of ketamine, approximately 24 hours apart, in the first four postpartum day
3. Receive additional therapy sessions before (to prepare for ketamine) and after (interpersonal therapy) each ketamine injection
4. Undergo assessments of brain electrical activity (at rest and evoked by trans-cranial magnetic stimulation) before and at three timepoints in the 10 hours after each ketamine injection
5. Complete mood assessments over the first 12 postpartum weeks

DETAILED DESCRIPTION:
The investigators will perform an open-label case series to evaluate the feasibility of performing a trial of a novel intervention to reduce postpartum depression symptoms after cesarean delivery. The intervention, Perinatal SMILES (Synergistic Multi-component Intervention to alLeviate dEpressive Symptoms), combines interpersonal therapy with subcutaneous ketamine therapy. The interpersonal therapy consists of five sessions that will be administered during the antepartum and/or postpartum. The ketamine therapy will be administered as two injections, approximately 24 hours apart, in the first four postpartum days and will be preceded and followed by additional therapy sessions. The investigators will assess brain electronic activity before and after the ketamine injections and mood in the first 12 postpartum weeks. The objective is to determine the feasibility of recruiting participant, administering the intervention and collect the outcome data.

ELIGIBILITY:
Inclusion Criteria

English-speaking (necessary for IPT under the limitations of the pilot) Socio-economically disadvantaged (i.e., low-income requiring public assistance) Suffering with depressive symptoms (EPDS > 10) >18 years of age > 20 weeks pregnant scheduled for cesarean delivery" or "within 48 hours of an unscheduled (or scheduled) cesarean delivery.

Exclusion Criteria

An allergy to ketamine

Contraindications for TMS including the presence of metallic objects within 30 cm of the TMS coil, intracranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed; presence of intracardiac lines, defibrillators or a cardiac pacemaker and unable to assess safety; presence of implanted electronic devices that control physiologic functions and unable to assess safety

Have a personal history of a primary seizure disorder or a seizure associated with an intracranial lesion

History of severe head trauma or neurological disorders (e.g., pre-eclampsia) that substantially increase seizure risk, per PI discretion

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be >20 weeks pregnant
Enrollment: 0 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | through postoperative day 84
  These will be assessed using the Edinburgh Postpartum Depression Scale (EDPS) questionnaire.30 The EPDS is a set of ten questions about the subject's mood in the previous seven days. Each symptom is scored on a numeric rating scale of none (0) to severe (3). Commonly employed thresholds for psychiatric referral are 10-13 out of a possible 30 points.
P30 (TMS-evoked potential) | 4 days
  This will be assessed using TMS-EEG. The amplitude of each of component positive (P) and negative (N) deflections in the evoked EEG signal will be recorded before and at 3 timepoints in the 2-10 hours after ketamine. The component deflections are named according to polarity of the deflection (N = negative, P = Positive) and the approximate time in milliseconds after the TMS input. For example N45 is the negative deflection observed approximately 45 ms after the TMS input.
N45 (TMS-evoked potential) | 4 days
  This will be assessed using TMS-EEG. The amplitude of each of component positive (P) and negative (N) deflections in the evoked EEG signal will be recorded before and at 3 timepoints in the 2-10 hours after ketamine. The component deflections are named according to polarity of the deflection (N = negative, P = Positive) and the approximate time in milliseconds after the TMS input. For example N45 is the negative deflection observed approximately 45 ms after the TMS input.
P60 (TMS-evoked potential) | 4 days
  This will be assessed using TMS-EEG. The amplitude of each of component positive (P) and negative (N) deflections in the evoked EEG signal will be recorded before and at 3 timepoints in the 2-10 hours after ketamine. The component deflections are named according to polarity of the deflection (N = negative, P = Positive) and the approximate time in milliseconds after the TMS input. For example N45 is the negative deflection observed approximately 45 ms after the TMS input.
N100 (TMS-evoked potential) | 4 days
  This will be assessed using TMS-EEG. The amplitude of each of component positive (P) and negative (N) deflections in the evoked EEG signal will be recorded before and at 3 timepoints in the 2-10 hours after ketamine. The component deflections are named according to polarity of the deflection (N = negative, P = Positive) and the approximate time in milliseconds after the TMS input. For example N45 is the negative deflection observed approximately 45 ms after the TMS input.
Cortical evoked activity (CEA) | 4 days
  The CEA will be calculated from the area under the curve of the rectified single pulse TMS-evoked potential
Anxiety | through postoperative day 84
  This will be assessed using the General Anxiety Disorder-7 (GAD-7) questionnaire. There are 7 items scored from 0-3. The total score can range from 0 (no anxiety) - 21 (most anxiety).
Psychosocial stress | at enrollment 1 day
  This will be assessed using the Antenatal Risk Questionnaire (ANRQ). The range of scores is 5-60. A higher score indicates greater psychosocial risk.
Post-Traumatic Stress Disorder (PTSD) | through postoperative day 84
  The Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) questionnaire. Scores range 0 - 80. More severe PTSD scores higher.
Obstetric Quality of Recovery | through postoperative day 84
  (ObsQoR10 score, 10 items, total score 0-100)
Number of participants who successfully breastfeed their newborn baby | 4 days
  Success in any 24-hour period will be defined as when an infant breastfeeds, for 10 minutes or more in a rhythmic suck/swallow/pause/suck pattern, at least eight times in that 24-hour period.
Adverse effects - sedation | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): sedation.
Adverse effects - Blurred vision | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): blurred vision.
Adverse effects - diplopia | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): diplopia.
Adverse effects - dizziness | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): dizziness.
Adverse effects - euphoria | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): euphoria.
Adverse effects - amnesia | 4 days
  Each of the following will be assessed on a four point scale (Not present, mild, moderate, severe): amnesia.
Adverse effects - hallucinations | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): hallucinations.
Adverse effects - nystamus | 4 days
  Will be assessed on a four point scale (Not present, mild, moderate, severe): nystagmus.
Antidepressant treatment | through postoperative day 84
  All current pharmacological and psychological therapies will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: David Monks, MBCHB, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No